CLINICAL TRIAL: NCT04416477
Title: Duration of Immunity 10 Years After a Dose-response Study With Yellow Fever Vaccine - Complementary Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 001/2019
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Yellow Fever Vaccine
Keywords: Immunity duration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A volume of up to 10 mL of whole blood should be collected without anticoagulant. There will be at most two attempts at blood collection per participant.
  The study samples will be aliquoted and after will be stored for a maximum of 10 years in the biorepository of the Institute of Technology in Immunobiologicals (Bio-Manguinhos), Fiocruz, Rio de Janeiro, Brazil, and this time will begin at the end of the last participant's collection.
  An additional written Informed Consent Form will assess whether the participant wishes to donate part of the samples to Bio-Manguinhos BioBank. In this case, the biological sample shall be stored for an indeterminate period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Yellow fever is an acute febrile infectious disease transmitted to man urban cycle by mosquitoes infected by an arbovirus of the genus Flavivirus family Flaviviridae. Its occurrence is recorded in South America Central America and Africa. In cities the yellow fever vector is the Aedes aegypti mosquito which also transmits dengue viruses zika and chikungunya. This disease is more frequent in males and the most affected age group is above fifteen years due to the greater exposure related to the penetration in wild areas of the endemic zone of yellow fever. Another risk group is unvaccinated people who live near wild environments where the virus circulates. According to the World Health Organization a single dose of the yellow fever vaccine is sufficient to maintain protective immunity against yellow fever for a lifetime therefore a booster dose is not required. This question is difficult to evaluate because there is no serological correlate of protection against yellow fever and seropositivity is defined with several cut off points. Although studies indicate that the duration of protection after vaccination is long there is considerable evidence in the literature that antibody titer falls over the years reaching levels considered as seronegative in at least a portion of the vaccinees. This is of more concern to people living in endemic areas who are exposed to the virus throughout their lives. For this reason Brazil recommended revaccinating once at least until additional studies were done. The need to increase Bio Manguinhos production capacity to meet the increased demand from Brazil and other countries is urgent. The occurrence of epidemics when millions of individuals need to be vaccinated in a short period of time exceeds production capacity and this is a recurrent problem. The current vaccine has a very high potency well above the thousand international units recommended by World Health Organization. But we need to generate additional evidence that very low doses of viral particles in the yellow fever vaccine are still immunogenic and that their immunogenicity can be maintained for at least ten years after vaccination. This evidence will support the rapid increase of their availability by the fractionation of doses or other alternatives.

DETAILED DESCRIPTION:
This is an observational study in young adult males who received the first dose of the yellow fever vaccine when they participated in the Dose response study of the yellow fever vaccine produced by Bio Manguinhos Fiocruz. The purpose of this study is to know whether reduced dose immunity is maintained for at least ten years. This information is crucial to support the recommendation to use fractional dose in adults a topic of great interest to World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* Have participated as a volunteer of the study carried out in 2009.
* Seronegative volunteers before vaccination in the study "Dose-response study of yellow fever vaccine 17DD produced by Bio-Manguinhos / Fiocruz" carried out in 2009. Non-revaccinated volunteers, seropositive in the study "Duration of immunity to yellow fever in volunteers eight years after a dose-response study", conducted in 2017.
* Not having received another yellow fever vaccine after participating in the study "Dose-response study of the yellow fever vaccine produced by Bio-Manguinhos / Fiocruz" carried out in 2009 and the study "Duration of immunity to yellow fever in volunteers eight years after a dose-response study", conducted in 2017.
* Available to follow up during the field study period.
* Agree to give name, address, phone, and other contact information, if necessary.
* Agree to strictly follow the study protocol.
* Able to understand and sign the Informed Consent Form (ICF).
* Understand the impossibility of participating in another clinical trial during the time of participation in this study.

Note: Individuals with a history of travel to areas endemic for yellow fever may be included but will be analyzed separately.

Exclusion Criteria:

* Refusal to collect biological material (blood).

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Participants will be healthy male adults who received the first dose of the yellow fever vaccine in 2009 when they participated in the "Dose-response study of the yellow fever vaccine 17DD produced by Bio-Manguinhos / Fiocruz".
  Participation in the study will be documented at the time of signing the Informed Consent Form.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of individuals who were protected 10 years after the first dose of the yellow fever vaccine, assessed by the neutralization test | 10 years after the first dose of yellow fever vaccine
  Serological status of yellow fever in adult individuals 10 years after seroconversion in a low dose or full dose study of the 17DD yellow fever vaccine produced by Bio-Manguinhos / Fiocruz.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Homma, Principal Investigator — Instituto de Tecnologia em Imunobiológicos Bio-Manguinhos / FIOCRUZ
Locations (1):
- Unidade de Ensaios Clínicos em Imunobiológicos / Instituto de Tecnologia em Imunobiológicos de Bio-Manguinhos / Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vianna CM, Noronha TG, Camacho LAB, Andrade RC, de Souza Brum RC, Dos Santos EM, Aguiar DF, Dos Santos MLB, de Souza Cruz RL, de Lima SMB, de Souza Azevedo Soares A, Schwarcz WD, da Matta de Castro T, Xavier JR, da Conceicao DA, Homma A, de Lourdes de Sousa Maia M. Duration of post-vaccination immunity to yellow fever in volunteers ten years after a dose-response study - A complementary study. Vaccine. 2024 Oct 24;42(24):126083. doi: 10.1016/j.vaccine.2024.06.050. Epub 2024 Jun 25. PMID 38926068